CLINICAL TRIAL: NCT01375062
Title: Isolation, Culture and Characterization Stem Cells From Testis Biopsy
Brief Title: Obtaining Undifferentiated Cells From Testis Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Igenomix (Industry)
Responsible Party: Principal Investigator, Carlos Simon, Principal Investigator; Gynecologist IVI Valencia, Instituto Valenciano de Infertilidad, IVI VALENCIA
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0902-057-F-CS
Record Dates: First submitted 2011-06-07; First posted 2011-06-17 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2014-03

CONDITIONS: Azoospermia
MeSH Terms: conditions — Azoospermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tissue from biopsies (No Intervention)
  Interventions: Other: analyse and proliferate the cells

INTERVENTIONS:
Other: analyse and proliferate the cells — 1. Obtention of excess tissue from testicular biopsies and maintained in 4ºC until procedures.
  2. Digestion of the biopsies through controlled enzymes
  3. Replication of the cells
  4. Selection undifferentiated cells
  5. Expansion of the purification cells population
  6. Characterization of the cell population
  7. Assessment of pluripotent and germinal cell potential.
  8. Possible maturation of the cells.

SUMMARY:
The purpose of this study is to isolate and culture stem cell from adult human testicular biopsies for future transplantation in fertility preservation.

DETAILED DESCRIPTION:
Testicular biopsies were obtained from azoospermic patients as part of their diagnosis and work-up after obtaining a signed informed consent. A portion of each sample was mechanically dissected in PBS with 1% Pen/Strep. For enzymatic digestion samples were incubated with 0.5g/ml Collagenase type 1A for 20min and TripLE Select for 15min at 37ºC on a shaker and then filtered with 30µm and centrifuged at 1,000rpm. The pellets were seeded and incubated in embryonic stem cell media (hESC) with glial cell line-derived neurotrophic factor (GDNF 4ng/mL) for 5-7 days at 37ºC (1st culture). To identify and isolate SSCs they were marked with CD49f antibody and FACS sorted. Positive cells were cultured in gelatine plates containing hESC media with leukaemia inhibitory factor (LIF1000U/mL) (2nd culture).

ELIGIBILITY:
Inclusion Criteria:

-azoospermic patients

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Assessment of potential germinal and pluripotent of the isolated cultures. | one month
  •The spermatogonial cells isolated from testicular biopsies of azoospermic patients will be matured in vitro for thegeneration of sperm for infertility treatment.
  * Undifferentiated cells of the testis biopsy will be characterized as degrees of plasticity for proof that they are capable of regeneration spermatogenesis.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Simon, MDPhD, Study Director — IVI Valencia; Marcia Riboldi, PhD, Principal Investigator — Fundación IVI
Locations (1):
- IVI Valencia, Valencia, Spain